CLINICAL TRIAL: NCT01853592
Title: A Pilot Dosing Study for Gadofosveset Trisodium (Ablavar) for Coronary Magnetic Resonance Angiography (MRA)
Brief Title: Gadofosveset Trisodium for Heart Imaging Studies
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 130098; 13-CC-0098
Record Dates: First submitted 2013-05-02; First posted 2013-05-15 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2016-12-13

CONDITIONS: Obstructive Coronary Artery Disease; Coronary Arteriosclerosis; Coronary Artery Disease (CAD)
Keywords: Gadolinium Contrast; Cardiac MRI; MRA; MRI; MRI Safety
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Magnetic resonance imaging (MRI) is type of imaging study that uses magnetic fields and radio waves to take pictures of the body. To help the images show up more clearly, a contrast agent is injected into a vein. Researchers are interested in finding contrast agents that can help show problems with the blood vessels around the heart. They want to test an agent called Gadofosveset Trisodium to see how it works in MRI scans.

Objectives:

- To test the effectiveness of Gadofosveset Trisodium as a contrast agent in heart MRI scans.

Eligibility:

- Healthy volunteers between 18 and 45 years of age.

Design:

* Participants will be screened with a physical exam and medical history. They will provide blood samples before the scanning sessions.
* Participants will have an MRI scan after the screening visit. They will have a dose of the contrast scan before the study.
* Participants will return for one additional MRI scan within 1 to 2 months of each scan. Different doses of the contrast agent will be used for each scan.
* An additional blood sample will be collected within 1 week of the second MRI scan.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the diagnostic quality of contrast-enhanced coronary magnetic resonance angiography (MRA) is improved by using a higher versus a lower dose of a gadolinium-based contrast agent. We will compare two doses of an intravascular contrast agent (Gadofosveset, 0.03 and 0.06 mmol/kg) in this pilot dosing study. Healthy participants will be recruited who do not have a clinical indication for MR angiography but do have safety clearance for IV gadolinium contrast and MR scanning.

Subjects will be evaluated in order to determine if the signal to noise ratio (SNR) and contrast to noise ratio (CNR) of the coronary arteries is increased for the higher dose contrast agent. Parameters will be compared with paired t-testing for significance.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Able to understand and sign informed consent.

B. Able to complete an MRI scan.

C. Age 18-45 years old.

D. eGFR greater than or equal to 60mL/min/1.73m(2) within 1 week prior to gadolinium injection.

E. NIH employees may be involved and NIH requirements will be followed as laid out in NIH Policy Manual 2300-630-3 - Leave Policy for NIH Employees Participating in NIH Medical Research Studies.

F. Willing to travel to the NIH for scheduled follow-up visits and scans as well as potential repeat scans in the event of sub-optimal scanning.

EXCLUSION CRITERIA:

Individuals will be excluded from the study if they have:

A. Contra-indications to undergoing a MRA

Please review Radiology MRI section MRI safety questionnaire.

B. MRI with contrast within the last 6 months (self-reported) outside of our protocol.

C. Contra indications to receiving gadolinium-based contrast agent (specified here and on MRI safety questionnaire):

1. Allergy to gadolinium-based contrast
2. Labs:

i. Kidney and liver function above the upper limits of normal

ii. eGFR < 60ml/min/1.73m(2)

iii. Pregnancy test: positive

c. Acute renal failure, renal transplantation, curent dialysis treatment or hepatorenal syndrome

d. History of liver transplantation or severe liver disease

e. Severe Asthma

f. Hemoglobinopathies

g. History of multiple myeloma

h. History of significant allergic reaction to gadolinium-based contrast agents

i. Evaluated to be at increased risk for Nephrogenic Systemic Fibrosis (NSF).

D. Current written (or self-reported) record of:

1. atrial fibrillation
2. cardiac surgery
3. cancer treatment
4. other comorbid conditions that otherwise indicates the participant has renal function that may deteriorate between study procedures due to the participant s underlying medical condition or that would not allow the study subject to complete the protocol.

E. Current written (or self-reported) record of active:

1. Clinically diagnosed angina, heart failure, and/or clinically significant electrical conduction abnormality in the heart.
2. Pregnancy or lactation
3. Mental, neurologic or social condition preventing understanding of the rationale, procedures, risks and potential benefits associated with the trial
4. Paralyzed hemidiaphragm
5. Over 400 lbs and/or a body circumference that prevents adequate MRI gantry insertion.
6. Unable to lay flat in the scanner
7. Claustrophobia otherwise requiring anesthesia or sedation to undergo MRI.
8. Participant is not able to undergo intravenous line placement and/or refuse gadolinium contrast.

F. Any other conditions that precludes safety for MRI per the researcher s evaluation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03-08; Primary Completion 2014-02-11 (Actual); Study Completion 2016-12-13 (Actual)

PRIMARY OUTCOMES:
To evaluate 0.06 mmol/kg Gadofosveset trisodium compared to 0.03 mmol/kg Gadofosveset trisodium for the diagnostic quality of MRA of the coronary arteries, as measured by changes in signal to noise & contrast to noise ratios. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: David A Bluemke, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rhee CM, Bhan I, Alexander EK, Brunelli SM. Association between iodinated contrast media exposure and incident hyperthyroidism and hypothyroidism. Arch Intern Med. 2012 Jan 23;172(2):153-9. doi: 10.1001/archinternmed.2011.677. PMID 22271121
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Gerber TC, Carr JJ, Arai AE, Dixon RL, Ferrari VA, Gomes AS, Heller GV, McCollough CH, McNitt-Gray MF, Mettler FA, Mieres JH, Morin RL, Yester MV. Ionizing radiation in cardiac imaging: a science advisory from the American Heart Association Committee on Cardiac Imaging of the Council on Clinical Cardiology and Committee on Cardiovascular Imaging and Intervention of the Council on Cardiovascular Radiology and Intervention. Circulation. 2009 Feb 24;119(7):1056-65. doi: 10.1161/CIRCULATIONAHA.108.191650. Epub 2009 Feb 2. No abstract available. PMID 19188512
- [Derived] Ahlman MA, Raman FS, Pang J, Zemrak F, Sandfort V, Penzak SR, Fan Z, Liu S, Li D, Bluemke DA. Part 2 - Coronary angiography with gadofosveset trisodium: a prospective intra-subject comparison for dose optimization for 100 % efficiency imaging. BMC Cardiovasc Disord. 2016 Mar 22;16:58. doi: 10.1186/s12872-015-0152-8. PMID 27004532